CLINICAL TRIAL: NCT03184727
Title: Pulmonary Vasculature and Right Heart Dysfunction in Chronic Obstructive Pulmonay Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Chief of Pulmonary Vascular Disease Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2016YFC1304405
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: COPD; Pulmonary Vascular Disorder; Right Ventricular Dysfunction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pulmonary vasculopathy and right heart dysfunction in COPD are drawing increasing attention these days. Recent researches show that pulmonary vasculopathy and right heart dysfunction relate to greater severity in COPD. Applying appropriate modalities for early detection of pulmonary vasculopathy and right heart dysfunction is of great importance. What's more, the interaction mechanism between pulmonary vasculature, right heart and COPD still needs to be further studied. The aim of our study is to develop an assessment system of pulmonary vasculopathy and right heart dysfunction in COPD patients and elucidate their impact on COPD course and outcome.

ELIGIBILITY:
Inclusion Criteria:

* stable COPD patients

Exclusion Criteria:

* patents with other respiratory diseases and pulmonary hypertension other than group 3 PH;
* psychopath, addict or patients not able to coordinate;
* patients in pregnancy or breastfeeding;
* patients with limited life expectancy;
* patients with contraindiction for MRI or PET;
* patients having cerebrovascular events in 3 months;
* unstable COPD patients

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: stable COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 3 years
  survival rate in %

SECONDARY OUTCOMES:
COPD exacerbations | 3 year
  total times
GOLD degree | 3 year
  Ⅰ-Ⅳ according to the pulmonary function
NYHA degree | 3 year
  Ⅰ-Ⅳ according to the symptom

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Institute and Fu Wai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided